CLINICAL TRIAL: NCT00210457
Title: Phase III, Multicentre, Open Study to Assess the Efficacy and Safety of Lanreotide Autogel (60, 90 or 120 mg) in Acromegalic Patients Previously Treated or Not by Somatostatin Analogues.
Brief Title: Efficacy and Safety of Lanreotide Autogel (60, 90 or 120 mg) in Acromegalic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-54-52030-081
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation)

SUMMARY:
To evaluate the long-term efficacy and safety of repeated injections of lanreotide Autogel given in doses titrated to effect in acromegalic patients previously treated or not with somatostatin analogues.

ELIGIBILITY:
Inclusion Criteria:

* Patient having documentation supporting diagnosis of active acromegaly in one of the following definitions:

  * patient having received neither somatostatin analogue nor dopaminergic agonist within the previous 12 weeks and having an IGF-1 level at least 1.3 times the upper limit of the age-adjusted normal range,
  * patient being treated with a somatostatin analogue (other than lanreotide autogel) or a dopaminergic agonist when attending the first visit and having at the end of the wash-out period an IGF-1 level at least 1.3 times the upper limit of the age-adjusted normal range.

Exclusion Criteria:

* Patient having had pituitary surgery within the previous 3 months
* Patient having received radiotherapy for acromegaly disease within the previous 36 months
* Patient being predicted to require pituitary surgery (adenomectomy) or receive radiotherapy during the study period
* Patient having received lanreotide autogel at any time before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2000-09; Primary Completion 2002-07-15 (Actual); Study Completion 2002-07-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having a normal (age-adjusted) serum insulin-like growth factor 1 (IGF-1) level at end point (Week 48)

SECONDARY OUTCOMES:
Percentage of variation from baseline of the IGF-1 levels expressed as a percentage of the upper limit of the age-adjusted normal range
Mean growth hormone (GH) levels
Number of patients having a serum GH level at or below 2.5ng/ml
Number of patients having a serum GH level at or below 1 ng/ml
Number of patients with no or reduced clinical signs of acromegaly
Long-term safety of repeated injections of lanreotide autogel at titrated doses

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (17):
- France (16):
  - Hôpital Sud, Amiens
  - Chu d'Angers, Angers
  - Hôpital de Bois Guillaume, Bois-Guillaume
  - Chu de la Cote de Nacre, Caen
  - Hôpital du Bocage, Dijon
  - Chu de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital du Cluzeau, Limoges
  - Hôpital Neurologique, Lyon
  - Hôpital Lapeyronie, Montpellier
  - Hôpital de l'Archet 1, Nice
  - Hôpital du Haut-Levêque, Pessac
  - Hôpital Maison Blanche, Reims
  - Hôpital Sud, Rennes
  - Hôpital Bellevue, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital de Rangueil, Toulouse
- Centre Hospitalier Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Chanson P, Borson-Chazot F, Kuhn JM, Blumberg J, Maisonobe P, Delemer B; Lanreotide Acromegaly Study Group. Control of IGF-I levels with titrated dosing of lanreotide Autogel over 48 weeks in patients with acromegaly. Clin Endocrinol (Oxf). 2008 Aug;69(2):299-305. doi: 10.1111/j.1365-2265.2008.03208.x. Epub 2008 Jan 31. PMID 18248639